CLINICAL TRIAL: NCT02029833
Title: Effects of Oleic Acid Enriched and Regular Canola Oil on Body Composition and Lipid Metabolism in Participants With Metabolic Syndrome
Brief Title: Canola Oil Multi-Centre Intervention Trial II
Acronym: COMIT2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Manitoba (Other)
Collaborators: Penn State University (Other); University of Toronto (Other); Laval University (Other); St. Boniface Hospital (Other); University at Buffalo (Other); Canola Council of Canada (Other); Agriculture and Agri-Food Canada (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: B2013:137
Record Dates: First submitted 2013-12-09; First posted 2014-01-08 (Estimated); Last update posted 2023-03-17 (Actual); Status verified 2021-04

CONDITIONS: Cardiovascular Disease; Diabetes; Metabolic Syndrome
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus; Metabolic Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Regular Canola Oil (Experimental): 60% oleic acid
  Interventions: Other: Regular Canola Oil
- High Oleic Canola Oil (Experimental): 70% oleic acid
  Interventions: Other: High Oleic Canola Oil
- Western Type Diet - Common Dietary Oils (Active Comparator): Ghee, Safflower oil, Coconut oil, & flax oil
  Interventions: Other: Western Type Diet - Common Dietary Oils

INTERVENTIONS:
Other: Regular Canola Oil
  Arms: Regular Canola Oil
Other: High Oleic Canola Oil
  Arms: High Oleic Canola Oil
Other: Western Type Diet - Common Dietary Oils
  Arms: Western Type Diet - Common Dietary Oils

SUMMARY:
The objectives of the study are to examine the health benefits of dietary canola oils on body composition, specifically on android fat, and weight management. COMIT II will also include analysis of FAEs to elucidate the mechanisms by which canola oil may be modifying body composition. Measurement of endothelial function, inflammatory, adiposity, and insulin sensitivity biomarkers will be done to determine the positive health impact of the changes in body composition achieved through canola oil consumption.

DETAILED DESCRIPTION:
The proposed multi-center clinical trial would engage the same collaborative team that successfully operationalized COMIT I, namely, the Richardson Centre for Functional Foods and Nutraceuticals (RCFFN) at the University of Manitoba (Winnipeg, Manitoba, Canada), the L'Institut Des Nutraceutiques et des Aliments Fonctionnels (INAF) at Laval University (Quebec City, Quebec, Canada), the Department of Nutritional Sciences at The Pennsylvania State University (University Park, Pennsylvania, USA), the Risk Factor Modification Centre at St. Michael's Hospital (Toronto, Ontario, Canada). St. Boniface Hospital Research (Winnipeg, Manitoba, Canada) will be an additional clinical trial site. The proposed COMIT II research program will proceed as a double blind, randomized crossover study consisting of three treatment phases of six weeks, each separated by a 6-week washout period. Participants will consume a fixed composition of a precisely controlled basal, weight-maintaining diet (35% energy from fat, 50% carbohydrate and 15% protein) supplemented with the following treatment oils: (a) regular canola oil, (b) high stability/ high oleic canola oil and (c) a typical "Western diet" fat intake as a control treatment comprised largely of saturated fat with substantial levels of omega-6 linoleic acid, common to current North American intakes. Treatment oils will be isocalorically incorporated into fruit smoothies made with milk and consumed at breakfast and supper. The clinical segment of COMIT II is expected to be completed by the mid to end of the second year, with sample analyses to be completed by the end of year three.

ELIGIBILITY:
Inclusion Criteria:

- Waist circumference ≥94 cm for men and ≥80 cm for women

Participants must meet at least one of the following secondary inclusion criteria:

* Fasting blood glucose of ≥ 5.6 mmol/L
* Triglycerides (TG) ≥1.7 mmol/L
* HDL cholesterol (HDL) <1 mmol/L (males) or <1.3 mmol/L (females)
* Blood pressure ≥130 mmHg (systolic) and/or ≥85 mmHg (diastolic).

Exclusion Criteria:

* Kidney, or liver disease, or unstable thyroid disease
* Diabetes mellitus
* Smokers
* Those consuming >1 alcoholic beverage a day for women and >2 for men.
* Any participant taking medication known to affect lipid metabolism or endothelial function

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 125 (Actual)
Dates: Start 2013-03; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Abdominal imaging of visceral and subcutaneous abdominal fat | 6 weeks
  Using a Dual Energy X-Ray Absorptiometry machine to analyze body composition, including measuring visceral adiposity. Units (fat mass) measured are cm3 and lbs.

SECONDARY OUTCOMES:
Analysis of fatty acid ethanolamides and precursors | 6 weeks
  Analysis of FAEs in the blood after consumption of treatment oils. UPLC-MS/MS will be used for FAE measurement.
Total lipid profiles including total cholesterol, high-density lipoprotein-cholesterol, low-density lipoprotein-cholesterol, triglyceride, and free fatty acid levels | 6 weeks
  Analysis of blood levels after consumption of treatment oils. Abbott Spectrum CCX Analyzer utilizing enzymatic reagents will be used to analyzed these measurements.
Plasma insulin level | 6 weeks
  Assessment of the change in insulin levels after consumption of treatment oils. This measurement will be analyzed by commercially available ELISA kits
Plasma glucose level | 6 weeks
  Assessment of changes in fasting glucose levels after consumption of treatment oils. This measurement will be analyzed by Abbott Spectrum CCX Analyzer
Plasma C-reactive protein level | 6 weeks
  Analysis of inflammatory marker levels after consumption of treatment oils will be conducted by ELISA kits
Plasma cytokines level | 6 weeks
  Analysis of inflammatory marker levels after consumption of treatment oils will be conducted by ELISA kits
Plant sterols and precursors of cholesterol | 6 weeks
  Analysis of plasma levels after consumption of treatment oils as indicators of cholesterol absorption and synthesis. These analysis will be conducted by gas chromatography
Proprotein convertase subtilisin/kexin type 9 (PCSK9) | 6 weeks
  PCSK9 will be measured as a surrogate marker of bile acid synthesis via Ultra Performance Liquid Chromatography-MS/MS
Endothelial function | 6 weeks
  Assessment of arterial wall resistance and arterial elasticity after consumption of treatment oils It will be assessed using flow mediated dilation
Fatty acid synthesis rates i.e. monounsaturated fatty acids and long chain polyunsaturated fatty acids | 6 weeks
  Heavy water enrichment of each fatty acid methyl ester after consumption of treatment oils will be measured using a gas chromatography with combustion isotope-ratio mass spectrometry
Single nucleotide polymorphisms in candidate genes related to body composition and fatty acid and FAE metabolism | 6 weeks
  Assessment of the potential influence of each SNP in an individual's response to consumption of treatment oils will be conducted using 7500 Fast Real-Time PCR System
Gene expression of candidate genes related to body composition and fatty acid and FAE metabolism | 6 weeks
  Assessment of levels of gene expression after consumption of treatment oils will be measured using real-time quantitative PCR
Activity Monitoring | 6 weeks
  Assessment of 24 hour physical activity including steps taken, raw acceleration, activity counts, energy expenditures, physical activity intensity, body position, and sleep/wake measurements after consumption of treatment oils will be measured using ActiGraph GT3X+ activity monitor
Lipocalin-2 | 6 weeks
  Fecal and serum lipocalin-2 will be analyzed for subgroup of participants using ELISA kit
Lipopolysaccharide (LPS) | 6 weeks
  Serum LPS will be analyzed for subgroup of participants using the LAL assay

CONTACTS AND LOCATIONS:
Overall Officials: Peter Jones, PhD, Principal Investigator — University of Manitoba
Locations (4):
- The Pennsylvania State University, University Park, Pennsylvania, United States
- Canada (3):
  - St Boniface Hospital Research, Winnipeg, Manitoba
  - Richardson Centre for Functional Foods and Nutraceuticals, University of Manitoba, Winnipeg, Manitoba
  - Institute of Nutrition and Functional Foods, Laval University, Québec, Quebec

REFERENCES:
- [Derived] Hammad SS, Eck P, Sihag J, Chen X, Connelly PW, Lamarche B, Couture P, Guay V, Maltais-Giguere J, West SG, Kris-Etherton PM, Bowen KJ, Jenkins DJA, Taylor CG, Perera D, Wilson A, Castillo S, Zahradka P, Jones PJH. Common Variants in Lipid Metabolism-Related Genes Associate with Fat Mass Changes in Response to Dietary Monounsaturated Fatty Acids in Adults with Abdominal Obesity. J Nutr. 2019 Oct 1;149(10):1749-1756. doi: 10.1093/jn/nxz136. PMID 31291447
- [Derived] Bowen KJ, Kris-Etherton PM, West SG, Fleming JA, Connelly PW, Lamarche B, Couture P, Jenkins DJA, Taylor CG, Zahradka P, Hammad SS, Sihag J, Chen X, Guay V, Maltais-Giguere J, Perera D, Wilson A, Juan SCS, Rempel J, Jones PJH. Diets Enriched with Conventional or High-Oleic Acid Canola Oils Lower Atherogenic Lipids and Lipoproteins Compared to a Diet with a Western Fatty Acid Profile in Adults with Central Adiposity. J Nutr. 2019 Mar 1;149(3):471-478. doi: 10.1093/jn/nxy307. PMID 30773586